CLINICAL TRIAL: NCT04666805
Title: Effect of Endocrine Therapy Duration on Clinical Outcome of Patients With Hormone Receptor-positive Intraductal Carcinoma of the Breast: A Multicenter, Retrospective, Real-world Study
Brief Title: Effect of Endocrine Therapy Duration on Clinical Outcome of Patients With HR+ Intraductal Carcinoma of the Breast
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Hospital of China Medical University (Other)
Collaborators: The First Hospital of Jilin University (Other); Second Hospital of Jilin University (Other); Jilin Provincial Tumor Hospital (Other); Affiliated Zhongshan Hospital of Dalian University (Other); The First Affiliated Hospital of Dalian Medical University (Other); China-Japan Union Hospital, Jilin University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); The Fifth People's Hospital of Shenyang (Unknown); General Hospital of Benxi Steel & Iron (Group) Co., Ltd (Unknown); Affiliated Hospital of Hebei University of Engineering (Unknown); Fourth People's Hospital of Shenyang (Other)
Responsible Party: Principal Investigator, Bo Chen, Professor, First Hospital of China Medical University
Other Study IDs: FirstHCMU_CB_001
Record Dates: First submitted 2020-12-04; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; hormone receptor; aromatase inhibitor; recurrence; metastasis
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Tamoxifen; Toremifene; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Drug Group: Endocrine therapy drugs include selective estrogen receptor modulators (Tamoxifen, Toremifene) and aromatase inhibitors (Anastrozole, Letrozole, Exemestane), which have been widely used in the adjuvant treatment of hormone receptor positive breast cancer.
  Interventions: Drug: Tamoxifen; Drug: Toremifene; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane

INTERVENTIONS:
Drug: Tamoxifen — 20 mg/d, oral administration
Drug: Toremifene — 60 mg/d, oral administration
Drug: Anastrozole — 1 tablet (1 mg) per day, oral administration
Drug: Letrozole — Adjuvant therapy with letrozole for 5 years or until the disease relapses. Patients who have received tamoxifen adjuvant therapy for 5 years should continue to take Letrozole until the disease relapses. The recommended dose of Letrozole tablets is one 2.5 mg tablet administered once a day, without regard to meals. For patients with advanced breast cancer, treatment with Letrozole should continue until tumor progression is confirmed. Patients with liver and/or renal dysfunction (creatinine clearance rate ≥ 10 mL/min) do not need to adjust the dosage.
Drug: Exemestane — The recommended dose of Exemestane for adult and older patients with early and advanced breast cancer is one 25 mg tablet administered orally once a day after a meal. After 2-3 years of tamoxifen treatment, patients with early breast cancer should continue to use Tamoxifen in the case of no recurrence or contralateral breast cancer, until the completion of 5-year sequential adjuvant therapy with tamoxifen and exemestane. Patients with advanced breast cancer should continue to take Exemestane until the tumor progresses.

SUMMARY:
This study will investigate the relationship between the endocrine therapy and the survival of patients with hormone receptor positive intraductal carcinoma of the breast, and the optimal duration of medication. This study will also analyze the risk factors of recurrence and metastasis of hormone receptor positive intraductal carcinoma of the breast and establish a prognosis model to further clarify the specific reasons for recurrence and metastasis, adverse reactions, and drug withdrawal in patients with hormone receptor positive intraductal carcinoma of the breast after endocrine therapy.

DETAILED DESCRIPTION:
Intraductal carcinoma of the breast accounts for 20% of newly diagnosed breast cancer. In addition to necessary surgical treatment, 5-year endocrine therapy is also essential for patients with hormone receptor positive ductal carcinoma of the breast. Commonly used drugs include selective estrogen receptor modulators (Tamoxifen, Toremifene) and aromatase inhibitors (Exemestane, Anastrozole, Letrozole). Although these drugs can effectively reduce the recurrence and metastasis of ductal carcinoma of the breast, the adverse reactions of the above drugs significantly reduce the quality of life and treatment compliance of the patients. Therefore, the choice of endocrine therapy for intraductal carcinoma of the breast has been widely discussed. Is it possible for de-escalation of endocrine treatment intensity to reduce adverse reactions and improve patient compliance? Recently, a phase 3 clinical trial found that compared with placebo group, the adverse reactions of Tamoxifen group treated with 5 mg/d (conventional dose 20 mg/d) Tamoxifen for 3 years had less adverse reactions and achieved significant efficacy. This study revealed the reliable efficacy and safety of Tamoxifen, a low-dose drug for treatment of hormone receptor positive intraductal carcinoma of the breast. However, little is reported on the reasonable duration of Aromatase inhibitors for endocrine therapy in patients with intraductal carcinoma of the breast.

This study will investigate the relationship between the endocrine therapy and the survival of patients with hormone receptor positive intraductal carcinoma of the breast, and the optimal duration of medication. This study will also analyze the risk factors of recurrence and metastasis of hormone receptor positive intraductal carcinoma of the breast and establish a prognosis model to further clarify the specific reasons for recurrence and metastasis, adverse reactions, and drug withdrawal in patients with hormone receptor positive intraductal carcinoma of the breast after endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* (1)Female patients aged ≥ 18 years and ≤ 85 years
* (2)The primary lesions and lymph nodes of the breast must meet all of the following conditions:

  1. Histologically confirmed intraductal carcinoma of the breast, accompanied by microinvasion, with the infiltration range ≤ 1 mm;
  2. Have received radical resection or breast conserving surgery;
  3. Patients who have received breast conserving surgery must undergo pathological examination to confirm there is no residual cancer tissue on the cutting edge and receive postoperative radiotherapy within the prescribed dose and range;
  4. No lymph node metastasis (including micrometastasis) is detected by postoperative pathological examination;
  5. Immuno
  6. Immunohistochemical staining results are positive for estrogen receptor (ER) or progesterone receptor (PR), which is defined as ER or PR immunoreactivity intensity ≥1+ or expression percentage ≥ 1%.
* (3)A volunteer to participate in the study and willing to cooperate with follow-up

Exclusion Criteria:

* (1)Patients with newly diagnosed metastatic breast cancer or other malignant tumors without breast intraductal carcinoma;
* (2) Patients who have other malignant tumors before the initial diagnosis of intraductal carcinoma of the breast
* (3) Patients who have received endocrine therapy with drugs including Toremifene, Tamoxifen, Anastrozole, Letrozole or Exemestane before the initial diagnosis of intraductal carcinoma of the breast
* (4) Patients who have a serious comorbidity or other comorbidities that interfere with the conduct of the study, or those who are considered not suitable for participation in this study

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: patients with hormone receptor-positive ductal carcinoma of the breast
Sampling Method: Probability Sample
Enrollment: 1354 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival up to 16 years | Time from the first disease-free day to the end of the last follow-up, assessed up to 16 years
  Disease-free survival refers to the time from the first disease-free day (i.e. the operation day) to the day at which relevant event occurs.
Invasive disease-free survival up to 16 years | Time from the first disease-free day to the end of the last follow-up, assessed up to 16 years
  Invasive disease-free survival refers to the time from the first disease-free day (i.e. the operation day) to the day at which intraductal carcinoma of the breast recurs. The recurrent diseases include ipsilateral or contralateral breast cancer, local and distant recurrence of breast cancer, and death due to any reason.
Distant disease-free survival up to 16 years | Time from the first disease-free day to the end of the last follow-up, assessed up to 16 years
  Distant disease-free survival refers to the time from the first disease-free day (i.e. the operation day) to the day at which distant metastasis occurs.

SECONDARY OUTCOMES:
Overall survival up to 16 years | Time from the first disease-free day to the end of the last follow-up, assessed up to 16 years
  Overall survival refers to the first disease-free day to the time of death caused by any reason.

OTHER OUTCOMES:
Adverse events of endocrine therapy up to 16 years | Time from the first disease-free day to the end of the last follow-up, assessed up to 16 years
  The incidence, nature, and severity of adverse events (including serious adverse events)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Chen, MD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided